CLINICAL TRIAL: NCT06303089
Title: Tobacco Exposure and Influencing Factors of Smoking Cessation Among Chronic Kidney Disease Patients: A Cross-Sectional Study.
Brief Title: Tobacco Exposure and Influencing Factors of Smoking Cessation Among Chronic Kidney Disease Patients
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, A.P., Sun Yat-sen University
Other Study IDs: zzwee-quit (CKD) 23152
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation
Keywords: Chronic kidney disease; Smoking cessation behavior; Cross-sectional study; Tobacco-related knowledge, attitudes, and practice; Tobacco exposure
MeSH Terms: conditions — Smoking Cessation; Renal Insufficiency, Chronic; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Questionnaires assessed Chronic Kidney Disease patients: Participants who met the inclusion criteria below will be invited to fill in tobacco exposure questionnaires, smokers will be invited to complete smoking cessation questionnaires set.
  1. Participants aged 18 years or older;
  2. Participants with a confirmed diagnosis of Chronic Kidney Disease;
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — Participants will be asked to respond to the demographic information sheet, characteristics of smoking sheet, tobacco-related knowledge, perceptions of tobacco harm. Smokers will be asked the history of smoking cessation sheet, the Fagerstrom Test of Nicotine Dependence, Smoking Self-efficacy Questionnaire, Cigarette Withdrawal Scale, Intention to Quit Smoking sheet, Motivation to Quit Smoking sheet, Alcohol Use Disorders Identification Test, and International Physical Activity Questionnaire.

SUMMARY:
The purpose of this study is to describe the tobacco exposure and characteristics of patients with Chronic Kidney Disease (CKD) who quit smoking, to identify patients' tobacco-related knowledge, attitude, and practice (KAP) and explore the influencing factors of smoking cessation.

DETAILED DESCRIPTION:
Participants will be invited to recall their smoking status and tobacco-related KAP. Smokers need to identify their smoking cessation behavior.

First part: participants need to finish the questionnaire, which includes the demographic information sheet, characteristics of smoking sheet, and tobacco-related KAP. Including (a) patients' knowledge of health risks of tobacco and tobacco-related diseases (the delphi method was used to construct this knowledge questionnaire); and (b) perceptions of tobacco harm.

Second part: smokers need to finish the questionnaire, which includes history of smoking cessation sheet, attitudes towards tobacco control smoking cessation, nicotine dependence sheet, tobacco withdrawal symptoms sheet, intention to quit smoking sheet, ability to quit smoking sheet, alcohol use disorders and physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years or older;
2. Participants with a confirmed diagnosis of Chronic Kidney Disease;
3. Participants were able to speak and read Chinese.;

Exclusion Criteria:

1. Participants who with psychiatric illness, disorders of consciousness, communication impairments, were unable to communicate effectively;
2. Participants who have acute and life-threatening exacerbations which require urgent treatment;
3. Patients who currently involved in other smoking cessation programs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Kidney Disease Patients
Sampling Method: Non-Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of current smokers | Baseline
  A true or false sheet in the questionnaire.
Abstinence rates | Baseline
  A true or false sheet in the questionnaire.

SECONDARY OUTCOMES:
Nicotine dependence | Baseline
  The Fagerstrom Test for Nicotine Dependence (FTND) was applied to assess nicotine dependence, which has a set of 6 items with an overall score ranging from 0-10. High dependence was defined as an FTND score ≥7; medium dependence, a score ranging from 4-6; low dependence, a score ranging from 0-3.
Perceptions of tobacco harm | Baseline
  Knowledge of health hazards of active and passive smoking was applied to assess perceptions of tobacco harm. The questionnaire has a set of 17 items which was developed according to the literature review content. Participants were asked to answer whether the knowledge about tobacco harm contained in the entry is correct: yes, no, or don't know. the higher percentages of correct responses to each item of the knowledge subscale means the better mastery of self-awareness of the hazard of smoking.
knowledge of tobacco-related diseases | Baseline
  Tobacco-related chronic kidney disease (CKD) was applied to assess knowledge of tobacco-related diseases. The questionnaire has a set of 23 items which was developed according to the literature review content (The delphi method was used to construct this knowledge level questionnaire). This questionnaire was categorized into three subscales, namely cigarette smoking increases the risk of CKD (15 items), e-cigarettes and nephrotoxicity (2 items) and health benefits of smoking cessation for patients with CKD (6 items), with the answer: know, know a little, do not know or not sure. Higher scores of both subscales indicate the greater mastery of knowledge of tobacco-related diseases.
Smoking related attitudes | Baseline
  Smoking Rationalization Beliefs (SRBs) refer to the relevant attitudes that smokers use to rationalize their smoking behavior and maintain their smoking status. The simplification of the scale with 8 items, each question use a five-point likert scale with 1 being 'strongly agree' and 5 being 'strongly disagree'. The higher the score was, the lower the SRBs.
Self-efficacy level | Baseline
  Smoking Self-Efficacy Questionnaire (SEQ-12) was applied to assess the self-efficacy level. The SEQ-12 is a self-report inventory consisting of 12 items measuring the confidence of current and exsmokers in their ability to abstain from smoking in high-risk situations. The instrument is intended to measure two dimensions: internal stimuli (6 items) and external stimuli (6 items). Responses were solicited with a five-point Likert scale ranging from 1=not at all sure to 5=absolutely sure, where greater values indicated that the respondent perceived greater confidence in resisting smoking in the context.
Withdrawal symptoms | Baseline
  The 9-item version of Minnesota Nicotine Withdrawal Scale (MNWS) was used for detection of withdrawal symptoms, which was revealed to have two domains of negative affect and insomnia and three individual items. Participants rated the symptoms by using a 5-point Likert-type (0=not present to 4=severe). Higher values of the MNWS indicate more severe nicotine withdrawal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified individual participant data will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.